CLINICAL TRIAL: NCT04252118
Title: Safety and Efficiency of Mesenchymal Stem Cell in Treating Pneumonia Patients Infected With COVID-19
Brief Title: Mesenchymal Stem Cell Treatment for Pneumonia Patients Infected With COVID-19
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing 302 Hospital (Other)
Collaborators: Innovative Precision Medicine Group (IPM), Hangzhou, China. (Unknown); Huoshenshan Hospital (Other); Tianjin Haihe Hospital (Other); Vcanbio Cell and Gene Engineering Corp., Ltd. (Industry); Shenzhen Third People's Hospital (Other); Fifth Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Fu-Sheng Wang, Head of Treatment and Research Center for Infectious Diseases, Principle Investigator, Clinical Professor, Beijing 302 Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020003D
Record Dates: First submitted 2020-01-27; First posted 2020-02-05 (Actual); Last update posted 2020-04-15 (Actual); Status verified 2020-04

CONDITIONS: COVID-19
Keywords: COVID-19; Safety; Efficiency; Cell Therapy; Mesenchymal stem cell
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MSCs Treatment Group (Experimental): Conventional treatment plus MSCs Participants will receive conventional treatment plus 3 times of MSCs(3.0*10E7 MSCs intravenously at Day 0, Day 3, Day 6).
  Interventions: Biological: MSCs
- Conventional Control Group (No Intervention): Without MSCs Therapy but conventional treatment should be received.

INTERVENTIONS:
Biological: MSCs — 3 times of MSCs(3.0*10E7 MSCs intravenously at Day 0, Day 3, Day 6).
  Arms: MSCs Treatment Group

SUMMARY:
The SARS-CoV-2 infection caused clusters of severe respiratory illness similar to severe acute respiratory syndrome coronavirus and was associated with ICU admission and high mortality. There is no confirmed antivirus therapy for people infected SARS-CoV-2, most of them should receive supportive care to help relieve symptoms. For severe cases, treatment should include care to support vital organ functions. This clinical trial is to inspect the safety and efficiency of Mesenchymal Stem Cells (MSCs) therapy for pneumonia patients infected with SARS-CoV-2.

DETAILED DESCRIPTION:
SARS-CoV-2 infection has become an urgent public health event in China. As of 24:00 on January 26, 2020, there are 2744 confirmed cases and 461 severe cases in China, the number is still increasing. There is currently no vaccine and no specific antiviral treatment recommended for SARS-CoV-2 infection. About 20% of the patients were severe and some died of respiratory failure or multiple organ failure. Therefore, it is urgent to find a safe and effective therapeutic approach to pneumonia patients infected with SARS-CoV-2.

In the last year, the promising features of mesenchymal stem cells (MSCs), including their regenerative properties and ability to differentiate into diverse cell lineages, have generated great interest among researchers whose work has offered intriguing perspectives on cell-based therapies for various diseases. These findings seem to highlight that the beneficial effect of MSC-based treatment could be principally due by the immunomodulation and regenerative potential of these cells. The investigators found that infusions of UC-MSC significantly improved liver function in decompensated liver cirrhosis and primary biliary cirrhosis (PBC) patients, increased the survival rate in acute-on-chronic liver failure (ACLF) patients . MSCs could significantly reduce the pathological changes of lung and inhibit the cell-mediated immune inflammatory response induced by influenza virus in animal model .

The purpose of this study is to investigate safety and efficiency of MSCs in treating pneumonia patients infected with SARS-CoV-2. This multi-center trial will recruit 20 patients. 10 patients received i.v. transfusion one round (3 times) of 3.0*10E7 cells of MSCs as the treated group, all of them received the conventional treatment. In addition, the equal 10 patients received conventional treatment were used as control. The clinical symptoms, pulmonary imaging, side effects, 28-days mortality, immunological characteristics (immune cells, inflammatory factors, etc.) will be evaluated during the 180 days follow up.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged at 18 years (including) -70 years old
2. Confirmed COVID-19 by reverse-transcription polymerase chain reaction (RT-PCR) from any diagnostic sampling source; and
3. Pneumonia that is judged by chest radiograph or computed tomography.

Exclusion Criteria:

1. Pregnancy, lactation and those who are not pregnant but do not take effective contraceptives measures;
2. Patients with malignant tumor, other serious systemic diseases and psychosis;
3. Patients who are participating in other clinical trials;
4. Inability to provide informed consent or to comply with test requirements.
5. Co-Infection of HIV, tuberculosis, influenza virus, adenovirus and other respiratory infection virus.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-01-27 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Size of lesion area by chest radiograph or CT | At Baseline , Day 3, Day 6, Day 10, Day 14, Day 21，Day 28
  Evaluation of Pneumonia Improvement
Side effects in the MSCs treatment group | At Baseline , Day 3, Day 6, Day 10, Day 14, Day 21, Day 28, Day 90 and Day 180
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0

SECONDARY OUTCOMES:
Improvement of Clinical symptoms including duration of fever and respiratory | At Baseline , Day 3, Day 6, Day 10, Day 14, Day 21, Day 28
  Evaluation of Pneumonia Improvement
Time of nucleic acid turning negative | At Baseline , Day 3, Day 6, Day 10, Day 14, Day 21, Day 28, Day 90 and Day 180
  Marker for COVID-19
Rate of mortality within 28-days | Day 28
  Marker for efficacy of treatment
CD4+ and CD8+ T celll count | At Baseline , Day 3, Day 6, Day 10, Day 14, Day 21, Day 28, Day 90 and Day 180
  Marker of Immunological function
Alanine aminotransferase | At Baseline , Day 3, Day 6, Day 10, Day 14, Day 21, Day 28, Day 90 and Day 180
  Markers of organ function
C-reactive protein | At Baseline , Day 3, Day 6, Day 10, Day 14, Day 21, Day 28, Day 90 and Day 180
  Markers of Infection
Creatine kinase | At Baseline , Day 3, Day 6, Day 10, Day 14, Day 21, Day 28, Day 90 and Day 180
  Markers of organ function

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing 302 Military Hospital of China, Beijing, China

IPD SHARING:
Plan to Share IPD: No